CLINICAL TRIAL: NCT02846623
Title: Atezolizumab (PD-L1 mAb) in Combination With Obinutuzumab and Venetoclax for Patients With Chronic Lymphocytic Leukemia and Richter Transformation
Brief Title: Atezolizumab, Obinutuzumab, and Venetoclax in Treating Patients With Chronic Lymphocytic Leukemia, Small Lymphocytic Lymphoma, or Relapsed or Refractory Richter Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1097; NCI-2017-00183 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-1097 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-07-22; First posted 2016-07-27 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia; Recurrent Transformed Chronic Lymphocytic Leukemia; Refractory Transformed Chronic Lymphocytic Leukemia; Richter Syndrome; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — atezolizumab; obinutuzumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (obinutuzumab, atezolizumab, venetoclax) (Experimental): Patients receive obinutuzumab IV over 4-6 hours on days 1, 2, 8, and 15 of cycle 1 and on day 1 of cycles 2-9 and atezolizumab IV over 30-60 minutes on days 3-4 of cycle 1 and on days 1-2 of cycles 2-9. Treatment repeats every 28 days for 9 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 3, patients also receive venetoclax PO on days 1-28. Treatment repeats every 28 days for 14 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Other: Laboratory Biomarker Analysis; Biological: Obinutuzumab; Drug: Venetoclax
- Cohort II (obinutuzumab, atezolizumab, venetoclax) (Experimental): Patients receive obinutuzumab intravenously IV over 4-6 hours on days 1, 2, 8, and 15 of cycle 1 and on day 1 of cycles 2-9 and atezolizumab IV over 30-60 minutes on days 3-4 of cycle 1 and on days 1-2 of cycles 2-9. Treatment repeats every 28 days for 9 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 2, patients receive venetoclax PO on days 1-28. Treatment repeats every 28 days for 25 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Other: Laboratory Biomarker Analysis; Biological: Obinutuzumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759; RO-5072759; RO5072759
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well atezolizumab, obinutuzumab, and venetoclax work in treating patients with chronic lymphocytic leukemia or small lymphocytic lymphoma or Richter syndrome that has come back (recurrent) or does not respond to treatment (refractory). Immunotherapy with monoclonal antibodies, such as atezolizumab and obinutuzumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as venetoclax, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving atezolizumab, obinutuzumab, and venetoclax may work better in treating patients with chronic lymphocytic leukemia, small lymphocytic lymphoma, or Richter syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of atezolizumab in combination with obinutuzumab and venetoclax in patients with chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL)/Richter transformation (RT).

SECONDARY OBJECTIVES:

I. To determine the safety of atezolizumab combined with obinutuzumab and venetoclax in patients with CLL/SLL/RT.

II. To determine overall response rate (ORR), complete response rate (CR), duration of response (DOR), and minimal residual disease (MRD) negative remission rate.

III. To determine the progression-free survival (PFS). IV. To determine the overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To determine immunological and molecular features, at baseline and/or that change with treatment, that correlate with outcomes in patients treated with atezolizumab combined with obinutuzumab and venetoclax.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients receive obinutuzumab intravenously (IV) over 4-6 hours on days 1, 2, 8, and 15 of cycle 1 and on day 1 of cycles 2-9 and atezolizumab IV over 30-60 minutes on days 3-4 of cycle 1 and on days 1-2 of cycles 2-9. Treatment repeats every 28 days for 9 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 3, patients also receive venetoclax orally (PO) on days 1-28. Treatment repeats every 28 days for 14 cycles in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients receive obinutuzumab intravenously IV over 4-6 hours on days 1, 2, 8, and 15 of cycle 1 and on day 1 of cycles 2-9 and atezolizumab IV over 30-60 minutes on days 3-4 of cycle 1 and on days 1-2 of cycles 2-9. Treatment repeats every 28 days for 9 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 2, patients receive venetoclax PO on days 1-28. Treatment repeats every 28 days for 25 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion:

1. Patients will have a diagnosis of CLL or SLL or RTand are: a) Cohort 1: Patients with treatment naïve CLL/SLL who meet IWCLL criteria for treatment or b) Cohort 2: RT (treatment-naïve or R/R)
2. Age >/= 18 years
3. Eastern Cooperative Oncology Group (ECOG) Performance Status </= 2
4. Patients must have adequate renal and hepatic function: -- Serum bilirubin </= 1.5 x upper limit of normal (ULN). For patients with Gilbert's disease, serum bilirubin up to </= 3 x ULN is allowed provided normal direct bilirubin. -- Serum creatinine </= 1.5 x ULN, -- Alanine aminotransferace (ALT) and aspartate aminotransferase (AST) </= 2.5 x ULN
5. Females of childbearing potential [A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (>/=12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)] must have a negative serum or urine beta human chorionic gonadotrophin (b-hCG) pregnancy test result within 14 days prior to the first dose of treatment and must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of <1% per year during the treatment period and for 6 months following the last dose of the study drugs. Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
6. #5 Continued - Males who have partners of childbearing potential must agree to use an effective contraceptive method such as a barrier method during the study and for 6 months following the last dose of study drugs. Males should also refrain from donating sperm.
7. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
8. Patients or their legally authorized representative must provide written informed consent

Exclusion:

1. Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or localized prostate cancer. If patients have another malignancy that was diagnosed/treated within the last 2 years, such patients may be enrolled if the likelihood of requiring systemic therapy for this other malignancy within 2 years is less than 10%, as determined by an expert in that particular malignancy at MD Anderson Cancer Center and after consultation with the Principal Investigator.
2. Prior treatment with CTLA-4, PD-1, PD-L1, or CD137 mAb, or venetoclax.
3. Any major surgery, radiotherapy, chemotherapy, biologic therapy, immunotherapy, experimental therapy, investigational therapy within 4 weeks prior to the first dose of the study drugs. Note: for patients on oral targeted therapies, a wash-out of 3 days from cycle 1 day 1 is acceptable.
4. Adverse events from prior anticancer therapy that have not resolved to Grade </= 1 except for alopecia
5. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 3 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
6. History of stroke or cerebral hemorrhage within 3 months
7. Patients who have uncontrolled hypertension (defined as sustained systolic blood pressure >/= 160 mmHg or diastolic >/= 100 mmHg)
8. Known evidence of active cerebral/meningeal CLL. Patients may have a history of central nervous system (CNS) leukemic involvement if definitively treated with prior therapy and no evidence of active disease at the time of registration (defined as >/= 2 consecutive spinal fluid assessments with no evidence of disease)
9. Active, uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia requiring steroid therapy (>10mg/day of prednisone or equivalent).
10. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis), with the following exceptions: Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
11. #10 Continued: a. Rash must cover < 10% of body surface area b. Disease is well controlled at baseline and requires only low-potency topical corticosteroids c. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.
12. Patients with organ allografts (such as renal transplant) are excluded
13. Patients who are on high-dose steroids (doses >10mg/day of prednisone or equivalent) or immune suppression medications. NOTE: Patients on high-dose steroids (doses >10mg/day of prednisone or equivalent) or immune suppression medications are eligible provided these drugs are discontinued at least 3 days prior to starting on the study drugs
14. Patients with uncontrolled active infection (viral, bacterial, and fungal) are not eligible
15. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
16. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
17. Current or chronic hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
18. Patient is pregnant or breast-feeding or intending to become pregnant during the course of the study or within 6 months after the last dose of the study drugs.
19. Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies or fusion proteins.
20. Patients may not receive other concurrent investigational agent, chemotherapy, radiotherapy, or immunotherapy for CLL. NOTE: Localized radiotherapy to an area not compromising bone marrow function does not apply
21. Received strong CYP3A inhibitors or strong CYP3A inducers within 7 days of starting venetoclax
22. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during the course of the study or within 5 months after the last dose of atezolizumab.
23. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2017-01-31 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) negative rate (Cohort I) | At end of cycle 9
  The Bayesian approach of Thall, Simon, Estey will be implemented for the toxicity and futility monitoring. Toxicity is defined as any grade 3 or higher non-hematological toxicity which is at least possibly related to the treatment. The MRD negative rate will be estimated along with the 95% credible interval for cohorts 1 and 2.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 1 year
  Will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Safety data will be summarized by category, severity and frequency. The proportion of patients with AEs will be estimated, along with the Bayesian 95% credible interval.
Best overall response | Up to 14 cycles (cohort 1) or 26 cycles (cohort 2)
  Will be estimated along with the 95% credible interval.
Complete response rate | Up to 1 year
  Summary statistics will be provided for continuous variables. Frequency tables will be used to summarize categorical variables.
Duration of response | Up to 1 year
  Summary statistics will be provided for continuous variables. Frequency tables will be used to summarize categorical variables.
Progression-free survival | Up to 1 year
  Kaplan-Meier method will be used.
Overall survival | Up to 1 year
  Kaplan-Meier method will be used.

OTHER OUTCOMES:
Change in immunological and molecular features | Baseline up to 1 year
  Will determine if the change in immunological and molecular features will correlate with patient outcomes and will be assessed through fitting linear or non-linear mixed effect models.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org